CLINICAL TRIAL: NCT05661123
Title: Effect of Modified Complete Decongestive Therapy on Lower Limbs Fibrosis Post Cellulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eva Magdy Bottros Nakhla, Physical therapist and Certified lymphedema therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lymphedema,fibrosis
Record Dates: First submitted 2022-11-27; First posted 2022-12-22 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Lower Limb Lymphedema; Fibrosis; Cellulitis of Leg
Keywords: Lymphedema; complete decongestive therapy; kinesio tape
MeSH Terms: conditions — Fibrosis; Lymphedema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- will receive kinesio tape in addition to complete decongestive therapy for 6 successive weeks. (Experimental): will receive Complete decongestive therapy in combination with kinesio tape
  Interventions: Other: Complete decongestive therapy
- will receive complete decongestive therapy for 6 successive weeks. (Other): Complete Decongestive Therapy(traditional physical therapy) that includes:
  1. Education.
  2. Skin care .
  3. Pneumatic compression device .
  4. Manual lymph draining .
  5. Multilayer short stretch compression bandages.
  6. Exercises.
  Interventions: Other: Complete decongestive therapy

INTERVENTIONS:
Other: Complete decongestive therapy — 1. Education.
  2. Skin care .
  3. Pneumatic compression device .
  4. Manual lymph draining .
  5. Multilayer short stretch compression bandages.
  6. Exercises.

SUMMARY:
this study will be designed to investigate the therapeutic benefits of kinesio tape in combination to complete decongestive therapy on limb volume , skin fibrosis, functional capacity ,ankle range of motion, lymphedema associated symptoms (pain, tightness, heaviness and hardness) and quality of life in patients with lower limbs fibrosis post cellulitis ,as well as finding out a physical therapy approach that has positive effect in treatment and care such cases which would enhance the physical therapy field.

DETAILED DESCRIPTION:
Lymphedema patient need a rehabilitative intervention in two phases : decongestion phase to reduce edema volume , improve the skin extensibility and provide him a better quality of life, followed by the maintenance phase to keep the outcomes. When we use the kinesio tape in addition to the complete decongestive therapy, the patient will experience a better improvement in the edema volume and the skin extensibility within a shorter period of time , a lesser number of sessions and a lower cost. So, the patient will have a better quality of life and could be a productive person in the society.

ELIGIBILITY:
Inclusion Criteria:

The patient will be according the following criteria:-

1. Males and females with Lower limb lymphedema Stage 2.
2. Age will range from45 to 55years old.
3. BMI <40 (kg/m2).
4. All patients will be clinically and medically stable when attending the study.
5. Patients free from any acute conditions.
6. Post cellulitis for at least 2 weeks.

Exclusion Criteria:

1. Unstable cardiovascular problems.
2. Altered mental status or poor cognition.
3. Lower limb ischemia (ABI ≤0.8).
4. Lower limb lymphedema stage 3&4.
5. Acute deep venous thrombosis.
6. Any acute infection.
7. Patients with orthopedic or neurological limitations to exercise.
8. Any lower limb acute ulcer or arterial wounds.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To assess limb volume | 6 weeks
  using Circumferential tape measurement to measure round measurements in cm at the beginning of the study then every 3 sessions
To assess skin extensibility | 6 weeks
  using tonometer at the beginning of the study and at last session after 6 weeks
To evaluate ankle range of motion | 6 weeks
  using digital goniometer at the ankle joint to assess the dorsi flexion degree at the beginning of the study and at the last session
To evaluate patient quality of life | 6 weeks
  using Lymphedema life impact scale in form of 18 questions every question' answer from 0 ( no symptoms) to 4 ( sever symptoms) at the beginning of the study and at the end of sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Al Sahel teaching hospital, Cairo, Egypt